CLINICAL TRIAL: NCT03282305
Title: Prospective Cohort Assessing the Prevalence and Progress of Non-alcoholic Fatty Liver Disease (NAFLD)/Non-alcoholic Steatohepatitis (NASH) in Chinese
Brief Title: Great China Fatter Liver Consortium (GC_FLC) Study to Assess the Progress of NAFLD/NASH in Chinese
Status: Not yet recruiting | Type: Observational
Sponsor: Great China Fatty Liver Consortium Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: NASH_GC-FLC01
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be stored for biomarkers analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a progressive liver disease ranging from simple steatosis to cirrhosis of the liver. Nonalcoholic fatty liver (NAFL) without substantial hepatocellular injury is thought to be relatively benign whereas nonalcoholic steatohepatitis (NASH) is characterized by hepatocyte steatosis, ballooning, inflammation and varying degrees of fibrosis from none to cirrhosis. NASH is strongly associated with insulin resistance and metabolic syndrome and thus is recognized as a major public health concern as the most prevalent liver disease.

Liver biopsy is the gold standard for a diagnosis of NASH. However, given the large population of patients at risk for NASH, liver biopsy is not a practical method for determining which patients may benefit from NASH therapy. Non-invasive methods to estimate inflammation and fibrosis are in clinical use, but there remains a dichotomy between gold standard inclusion criteria and end points that are utilized in clinical trials and real world diagnostic methods that are more common in clinical practice.

Thus, the investigators would like to conduct an observational study to head-to-head compare the non-invasive methods and liver biopsy in differential liver steatosis and liver biopsy in a real-world setting. Also, by following up patients for a relatively long time (proposed 10 years), the investigators can present the natural history of disease progression.

DETAILED DESCRIPTION:
GC-FLC is a cooperative consortium of principal investigators from academic institutions and community-based sites treating patients with NAFLD and NASH. The investigators will leverage the multidisciplinary expertise within this network in bio-banking, high-throughput technologies, and biomedical informatics to give investigators the power to analyze effectiveness data at many different levels of resolution, ranging from subsets of patients to very large populations.

GC-FLC will use standardized data collection practices, study data monitoring, and an comprehensive observational protocol in order to increase the efficiency and minimize costs associated with performing clinical research while ensuring collection of detailed critical safety and effectiveness data on prescribed NASH therapies. GC-FLC engages community and academic practice providers as partners in the research to ensure rapid translation of research findings into improvement in healthcare quality and outcomes and to help engage scientists at the interfaces between clinical research and the community. Furthermore, GC-FLC provides the opportunity to pair-comparison between liver biopsy and non-invasive biomarkers in differential low-risk and high-risk population for treatment in real world settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children subjects aged >= 6 years old
* Ability to understand and sign a written informed consent form (ICF) or provide assent in pediatric subjects
* Diagnosis of NAFLD; or a definite or probable diagnosis of NASH:

  1. A diagnosis of NAFLD will be defined by evidence of hepatic steatosis, either by imaging or by histology, with no causes for secondary hepatic fat accumulation such as significant alcohol consumption, use of steato-genic medication (e.g. valproate, amiodarone, anti-retroviral medications, tetracycline, chronic high-dose corticosteroids), or hereditary disorders (e.g. Wilson's disease, Wolman disease, cholesteryl-ester storage disease);
  2. A definite diagnosis of NASH will be defined by steatohepatitis confirmed by biopsy with correlating clinical evidence of non-alcoholic liver disease;
  3. A probable diagnosis of NASH will be defined by:

     a.Elevated alanine amino transferase levels (ALT) of >40 U/L; and b.Evidence of hepatic steatosis on imaging; or c.Obesity, type 2 diabetes, or pre-diabetes. Pre-diabetes is defined by: i.Impaired fasting glucose: 100 mg/dL-125 mg/dL (5.6 mmol/L-6.9 mmol/L) or; ii.Impaired glucose tolerance: 2-hr plasma glucose (PG) in 75-g Oral Glucose Tolerance Test (OGTT) 140 mg/dL-199 mg/dL (7.8 mmol/L-11.0 mmol/L) or; iii.HbA1C: 5.7%-6.4%.

     Exclusion Criteria:
* Unable to provide written informed consent (or assent in pediatric subjects)
* Alcohol consumption greater than 21 units/week for males or 14 units/week for females (one unit of alcohol is half pint of beer [285 mL; 9.64 oz], 1 glass of spirits [25 mL; 0.85 oz] or 1 glass of wine [125 mL; 4.23 oz]
* Enrolled in NASH-related clinical trials
* Presence of other forms of chronic liver disease:

  1. Chronic hepatitis B (HBsAg positive)
  2. Chronic hepatitis C (HCV RNA positive)
  3. Iron overload disorders (3-4+ iron on liver biopsy or known hemochromatosis gene (HFE) C282Y homozygous with ferritin > 200 ng/ml; note: an elevated ferritin alone is common in NASH and is not exclusionary)
  4. Autoimmune liver disease (biopsy evidence or clinical diagnosis of autoimmune hepatitis or Primary biliary cholangitis (PBC) requiring ongoing treatment, imaging evidence of Primary sclerosing cholangitis (PSC))
  5. Wilson's disease
  6. Alpha-1 antitrypsin mutations that in the opinion of the principal investigator is contributing to the patient's liver disease;
* Prior bariatric surgery unless the surgery was performed more than one year before the biopsy diagnosis of NASH (i.e., NASH is present despite prior bariatric surgery);
* Planned bariatric surgery (e.g. gastroplasty, roux-en-Y gastric bypass).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese subjects with NAFLD / NASH
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Histological endpoint | 10 years
  The change in NASH Clinical Research Network (CRN) score based on liver biopsy

SECONDARY OUTCOMES:
Number of all-cause death | 10 years
  Number of all-cause death
Number of liver-related death | 10 years
  Number of liver-related death
Number of liver transplant | 10 years
  Number of liver transplant
Number of hepatocellular carcinoma (HCC) | 10 years
  Number of hepatocellular carcinoma (HCC)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Wong, MD, PhD, Principal Investigator — Department of Medicine & Therapeutics, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong SAR, China.; George Lau, MD, PhD, Study Chair — Division of Gastroenterology & Hepatology, Humanity & Health Medical Centre, Hong Kong SAR, China.; Arun Sanyal, MD, PhD, Study Director — Physiology and Molecular Pathology, School of Medicine, Virginia Commonwealth University, Richmond, Virginia, USA